CLINICAL TRIAL: NCT03973099
Title: Double Blinded, Randomized, Placebo-controlled Clinical Study for Evaluating Anti-stress Effects of Nelumbinis Semen by 2 Week Administration
Brief Title: Double Blinded, Randomized, Placebo-controlled Clinical Study for Nelumbinis Semen
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VTBIO Co. LTD (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KCMC07OT066
Record Dates: First submitted 2019-05-29; First posted 2019-06-04 (Actual); Last update posted 2019-06-04 (Actual); Status verified 2019-06

CONDITIONS: Stress
MeSH Terms: interventions — Nelumbinis Semen

STUDY DESIGN:
Intervention Model Description: Double blinded, randomized, placebo-controlled clinical study for evaluating anti-stress effects of Nelumbinis Semen
Who Masked: Participant, Investigator
Masking Description: Double-blind study : Participants and investigators do not know which treatment is placebo or treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Experimental): Subjects in the placebo group received the equivalent amount of starch and lactose mixture capsules and administered with the same schedule.
  Interventions: Dietary Supplement: PM011
- PM011 (Experimental): PM011 is a 400 mg hard gelatin capsule containing water extracts of Nelumbinis Semen. The sprayed-dry extract of the herbal medicine used was purchased from Sun Ten pharmaceutical company in Taiwan. Each participant received twelve capsules of PM011, which divided into 2.4 g treatment or 4.8 g treatment group or placebo daily for two weeks and was instructed to take six capsules after breakfast and six capsules after dinner.
  Interventions: Dietary Supplement: PM011

INTERVENTIONS:
Dietary Supplement: PM011 — PM011 is a 400 mg hard gelatin capsule containing water extracts of Nelumbinis Semen. The sprayed-dry extract of the herbal medicine used was purchased from Sun Ten pharmaceutical company in Taiwan. Each participant received twelve capsules of PM011, which divided into 2.4 g treatment or 4.8 g treatment group or placebo daily for two weeks and was instructed to take six capsules after breakfast and six capsules after dinner. Subjects in the placebo group received the equivalent amount of starch and lactose mixture capsules and administered with the same schedule.
  Other Names: Nelumbinis Semen

SUMMARY:
Nelumbinis Semen, has been widely used as treatment of post-menopause symptoms in women for hundreds of years in many Asian countries. This study examines whether PM011, standardized herbal medicine made from Nelumbinis Semen, treats stress in above 5 of BDI score of human subjects and discusses its potential as treatment for depressed patients.

DETAILED DESCRIPTION:
Nelumbinis Semen, has been widely used as treatment of post-menopause symptoms in women for hundreds of years in many Asian countries. This study examines whether PM011, standardized herbal medicine made from Nelumbinis Semen, treats stress in above 5 of BDI score of human subjects and discusses its potential as treatment for depressed patients. Subjects were divided into three groups, the placebo-treated group (n = 10), the PM011-2.4 g treated group (n = 11) and PM011-4.8 g treated group (n = 11) per day. Alpha/Beta ratio of electroencephalogram (EGG), Beck Depression Inventory (BDI) and Stress Response Inventory (SRI) were conducted in order to measure changes in stress before and after 2 weeks of PM011 treatment.

ELIGIBILITY:
<Inclusion Criteria>

* Volunteers were selected based on following meet conditions;Men and women, who have willingness and capacity to comply with the study protocol, are included if they were aged 18 to 65 years.
* Volunteers, who can understand Korean and English alphabet are selected.
* Volunteers, who can communicate with clinical trial performer fully, comply with the all tests and medical examinations performed by study protocol.
* All volunteers or their protectors understand purpose of study fully and sign their names or seal.
* Volunteers, who do not come under exclusion criteria are selected.
* BDI score of Volunteers, who can be >= 5.

<Exclusion Criteria>

* Volunteers were excluded if they are applied to following meet conditions; Volunteers with fasting glucose level over 126 mg/dl.
* Volunteers with hypertension as having over 140 mmHg of systolic blood pressure or 90 mmHg of diastolic blood pressure.
* Volunteers with blood thyroid stimulating hormone below 0.3 or over 4.0.
* Men with hemoglobin below 13.0 g/dl and women with hemoglobin below 12.0 g/dl.
* Volunteers with abnormality of liver function as having over 1.5 times of normal levels of ALT or AST.
* Patients with infections in upper airways or chronic diseases.
* Mental illness patients with such as alcoholism.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2007-06-07 (Actual); Primary Completion 2007-12-30 (Actual); Study Completion 2007-12-30 (Actual)

PRIMARY OUTCOMES:
Beck Depression Inventory (BDI) | Change from baseline BDI score at 2 weeks
  BDI is a 21 item, self rated inventory with each item rated with a set of four possible answer choices of increasing intensity.
Stress Response Inventory or Test (SRI or SRT) | Change from baseline SRI or SRT score at 2 weeks
  SRI is highly reliable and valid, and that it is utilized as an effective measure of stress for research in stress-related fields in Korea. SRI is a total of 39 response items under the seven subscales. The seven subscales are divided into tension (A), aggression (B), somatization (C), anger (D), depression (E), fatigue (F), and frustration (G). When the test is scored, a value of 0 to 4 is assigned for each answer and then the total score is compared to a key to determine the stress's severity.

SECONDARY OUTCOMES:
Alpha/beta ratio of electroencephalogram (EEG) | Change from baseline Alpha/beta ratio of electroencephalogram (EEG) at 2 weeks
  Electroencephalogram (EEG) is used to measure the brain waves. Each wave pattern is associated with different mood state and state of consciousness. Alpha is one of four basic brain waves (delta, theta, alpha and beta) which make up the EEG. Alpha is seen in wakefulness where there is relaxed and effortless alertness. Beta is seen in highly stressful situations, and where there is difficult mental concentration and focus. Therefore, high alpha and less beta waves have been used as indices of relaxation, arousal, anti-stress, and better concentration.

IPD SHARING:
Plan to Share IPD: No